CLINICAL TRIAL: NCT03381027
Title: BABY SMART (Study of Massage Therapy, Sleep And neurodevelopMenT)
Acronym: BabySMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Professor Geraldine Boylan, Professor Geraldine Boylan INFANT Centre Director, University College Cork
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GB02/17UCC
Record Dates: First submitted 2017-12-11; First posted 2017-12-21 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Sleep; Neurodevelopmental Disorders
Keywords: Infant Sleep; Baby Massage; Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: single centre, unblinded, randomised, controlled study to evaluate whether a multi-sensory enrichment programme in the first 4 months of life will improve sleep architecture and neurodevelopment in healthy infants.
Who Masked: Outcomes Assessor
Masking Description: Neurodevelopmental assessors are blinded to interventional arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm- Baby Massage (Experimental): Interventional Arm= Baby Massage
  Interventions: Procedure: Baby Massage
- Control Arm- no Baby Massage (No Intervention): Control Arm= no Baby Massage

INTERVENTIONS:
Procedure: Baby Massage — Structured massage of the baby
  Arms: Interventional Arm- Baby Massage

SUMMARY:
It is well known that sleep is essential for brain development and learning. Infants require extensive sleep for development of the hippocampus, pons, brainstem, and midbrain and for optimizing physical growth. It is also essential for brain plasticity; the genetically determined ability of the infant brain to change its structure and function in response to the environment. Studies in young animals have shown that sleep deprivation leads to increased programmed cell death, smaller brain size, and loss of brain plasticity, all of which have negative long-term impact on behaviour and learning ability.

Infant massage, a form of systematic tactile stimulation by human hands, improves sleep hygiene. Very little is known about how massage influences early brain development but it is certainly linked to the theory of environmental enrichment, which has been well established in animal models.

The aim of this project is to optimise the infant's sensory experience through a multi-sensory enrichment programme, including massage (a massage utilising a scented lotion before sleep each day), to encourage more structured sleep and ultimately show improved developmental and cognitive outcomes.

DETAILED DESCRIPTION:
See study protocol attached.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born > 37 weeks gestation
2. Single births
3. Not requiring admission to the Neonatal Unit
4. Healthy infants without suspected congenital or metabolic anomalies

Exclusion Criteria:

1. Infants born < 37 weeks gestation
2. Multiple births
3. Severe metabolic or genetic anomaly that would require ongoing specialist care in the infancy period.

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 408 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Infant sleep measured by video EEG length of sleep cycles | assessment carried out in fourth month of life
  Sleep EEG

SECONDARY OUTCOMES:
Neuro-development measured by Griffiths 3 Developmental Assessment | Assessment carried out at 4 & 18 month of life
  Griffiths 3 Developmental Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Boylan, PhD, Principal Investigator — INFANT UCC
Locations (1):
- Cork University Maternity Hospital, Cork, Munster, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] O Sullivan MP, Livingstone V, Korotchikova I, Dempsey EM, Murray DM, Boylan GB. Reference centiles for infant sleep parameters from 4 to 16 weeks of age: findings from an Irish cohort. Arch Dis Child. 2023 Jun;108(6):481-485. doi: 10.1136/archdischild-2022-324016. Epub 2023 Mar 21. PMID 36944485
- [Derived] Ventura S, Mathieson SR, O'Toole JM, Livingstone V, Ryan MA, Boylan GB. Electroencephalographic sleep macrostructure and sleep spindles in early infancy. Sleep. 2022 Jan 11;45(1):zsab262. doi: 10.1093/sleep/zsab262. PMID 34755881

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT03381027/Prot_SAP_000.pdf